CLINICAL TRIAL: NCT06595524
Title: Development of the Online Mindfulness-based Intervention (MFU-Mindful Application) for Thai-university Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University (Other)
Responsible Party: Principal Investigator, Chuntana Reangsing, Principle Investigator, Mae Fah Luang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Mae Fah Luang Unviersity
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depression in Adolescence; Psychological Well-Being
Keywords: depression; mindfulness; psychological well being; university students
MeSH Terms: conditions — Psychological Well-Being; Depression

STUDY DESIGN:
Intervention Model Description: Phase I: one group pre-posttest Phase II: randomized control trial
Who Masked: Outcomes Assessor
Masking Description: collecting all outcomes at baseline and post-intervention by using online web-based method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online mindfulness -base intervention (Experimental)
  Interventions: Behavioral: online mindfulness-based intervention
- waitlist control group (No Intervention)

INTERVENTIONS:
Behavioral: online mindfulness-based intervention — The mindfulness-based intervention (MFU-Mindful-application) consists of 8 topics, one topic per week. Moreover, we will assign participants (experimental group) to continuously practice using guided meditation approximately 10 minutes daily at least 5 days a week for 3 months via MFU-Mindful application
  Arms: online mindfulness -base intervention

SUMMARY:
Development of the online mindfulness-based intervention (MFU-mindful application) for Thai university students: Phase I

Objectives:

Phase I: (October 2021 to September 2022)

1. To develop the mindfulness-based intervention (MFU-Mindful application) for Thai university students.
2. To test the feasibility of the mindfulness-based intervention (MFU-Mindful Application) for Thai university students.
3. To determine the effect size of mindfulness-based intervention (MFU-Mindful Application) on mental health outcomes for Thai university students: A pilot study.

Phase II: (October 2022 to December 2024)

1. To examine the effects of mindfulness-base intervention (MFU-Mindful Application) on mental health outcomes for Thai university students

For this research project, investigators will develop the mindfulness-based intervention (MFU-Mindful application) based on mindfulness-based stress reduction (MBSR) and mindfulness-based cognitive therapy (MBCT) by encouraging participants to pay attention to their present thoughts, emotions, feelings, and behaviors without judgment. This attention will help them learn the relationship between their thoughts, emotions, and behaviors and their mental health outcomes (mindfulness, stress, anxiety, and depression) though mindfulness practice (body scan, sitting meditation, and mindful movement using online application). Also, investigators will teach participants how to shape their thoughts and manage their wondering minds and negative and irritable thoughts. Finally, participants will learn how to become an individual with reasonable, flexibility, and positive thoughts.

Population and sample:

Population: Thai university students who are between years 1-4 (undergraduate).

Sample:

Phase I: Mae Fah Luang University students who are studying during the Spring semester, year 2021. We will specifically recruit volunteers who:

Inclusion criteria:

1. are current studying in years 1-4 of undergraduate programs
2. can read, speak, and write in Thai
3. be risk of the mental health problem (score higher than 6 on the General Health Questionnaire (GHQ-28))
4. have no history of learning disorders (ADHD, other specific learning disorders)
5. have no psychiatric disorders (schizophrenia, adjustment disorders, delusion disorders, and substance use disorders)
6. have no meditation experience within the past 6 months

Exclusion criteria:

1. have a limitation for mindful movement (hearing loss, blindness, and movement limitations)
2. uncomfortable or feel distress and cannot participate in each mindful-based intervention session.

ELIGIBILITY:
We will specifically recruit volunteers who:

Inclusion Criteria:

1. are current studying in years 1-4 of undergraduate programs
2. can read, speak, and write in Thai
3. be risk of the mental health problem (score higher than 6 on the General Health Questionnaire (GHQ-28))
4. have no history of learning disorders (ADHD, other specific learning disorders)
5. have no psychiatric disorders (schizophrenia, adjustment disorders, delusion disorders, and substance use disorders)
6. have no meditation experience within the past 6 months

Exclusion Criteria:

1. have a limitation for mindful movement (hearing loss, blindness, and movement limitations)
2. uncomfortable or feel distress and cannot participate in each mindful-based intervention session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Suanprung Stress Test-20, SPST-20 | baseline-at week 8 (over 8 week)
  This is a self-administered questionnaire consisting of 20 items, which was adapted and translated into Thai by Mahatnirunkul et al. (1997). This scale provides one score reflecting sensitivity to stress, sources of stress, and physiological reactions to stress (e.g., muscular stress, nervous systems, emotional stress, and cognitive stress). This scale measures how much daily activities produce work-related stress and individuals' responses to stress. Respondents are asked to choose from five possible responses in a format requiring them to describe how they feel at this very moment on a 5-point intensity scale: 1 = no stress, 2 = mild stress, 3, = moderate stress, 4 = much stress, and 5=extreme stress. Higher scores indicate higher levels of stress. Researchers have divided the SPST-20 stress scores into four levels: 0-24, mild; 25-42, moderate; 43-62, high; and over 63, severe stress (Mahatnirunkul et al., 1997). Cronbach's alpha was reported to be more than .7 (Jitvaropas et al., 2
State-Trait Anxiety Inventory Form Y-1 | baseline- at week 8 (over 8 week)
  STAI form -1, Thai version. This scale is a self-report questionnaire developed by Spielberger and Sydeman (1994) and was translated into Thai by Thapinta (1991). This scale consists of 20 items including 10-positive items and 10-negative items. Respondents are asked to choose from four possible responses in a format requiring them to describe how they feel at this very moment on a 4-point intensity scale: 1 = not at all, 2 = somewhat, 3, = moderately, 4 = very much. Thus, possible scores ranged from 1 to 80. Higher scores indicate higher anxiety (Thapinta, 1991). For this study, the Cronbach's alpha coefficient was .80.
Philadelphia Mindfulness Scale, Thai version | baseline- at week 8 (over 8 week)
  This scale is a self-report questionnaire with 20 items, which was developed and translated by Silpakit et al. (2004). It consists of 2 subscales, awareness and acceptance, with response options from 1 to 5 (1=never, 2=rarely, 3=sometimes, 4=often, and 5=very often). A higher score indicates a higher mindfulness level. The Cronbach's alpha coefficient of awareness and acceptance among Thai-population were .87 and .88, respectively (Silpakit et al., 2004). For this study, the Cronbach's alpha coefficient was 0.92 for the total score.
Center for Epidemiologic Studies-Depression Scale-Thai version, CES-D-Thai version. | baseline- over 8 week
  CES-D Thai version is a self-report questionnaire with a total of 20 items, which was developed by the Center for Epidemiologic Studies at the U.S. National Institute of Mental Health and was translated and adapted into Thai by Trangkasombat et al. (1997). The reliability of this instrument was .86 among Thai adolescents (Trangkasombat et al., 1997). Respondents are asked to choose from four possible responses where 0 = rarely or none of the time (less than 1 day), and 4 = almost or all of the time (5 to 7 days). A total score is calculated by summing all items providing a possible range from 0 to 60. Higher scores reflect greater levels of depressive symptoms. The CES-D has 4 separate subscales: positive affect, negative affect, somatic symptoms, and interpersonal relations. Items on the positive affect subscale are reversed to reflect 'unhappy' or 'lack of well-being' (Trangkasombat et al., 1997). The CES-D has good internal consistency with alphas of 0.85 for the general population

CONTACTS AND LOCATIONS:
Locations (1):
- Mae Fah Luang University, Chiang Rai, Chiangrai, Thailand

IPD SHARING:
Plan to Share IPD: No
Prohibited from law